CLINICAL TRIAL: NCT02669225
Title: Characterization of Brain Amyloid-beta (A-beta) Retention During Wakefulness And Following Emergence From Sleep In Healthy Subjects
Brief Title: Brain Amyloid- Retention During Wakefulness and Following Emergence From Sleep in Healthy People
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 160059; 16-AA-0059
Record Dates: First submitted 2016-01-29; First posted 2016-02-01 (Estimated); Last update posted 2025-12-31 (Actual); Status verified 2025-10-22

CONDITIONS: Normal Physiology
Keywords: [18F]florbetaben; Sleep Deprivation; rested wakefulness; glymphatic system
MeSH Terms: conditions — Sleep Deprivation | interventions — 4-(N-methylamino)-4'-(2-(2-(2-fluoroethoxy)ethoxy)ethoxy)stilbene

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rested Wakefulness (Experimental): RW PET/MR Scanning Sessions
  Interventions: Other: [18F]florbetaben
- Sleep Deprivation (Experimental): SD PET/MR Scanning Sessions
  Interventions: Other: [18F]florbetaben

INTERVENTIONS:
Other: [18F]florbetaben — PET radiotracer to image Amyloid beta (AB) load in human brain.

SUMMARY:
Background:

Brain activity creates waste products. The body s glymphatic system removes this waste, especially during sleep. One brain waste product is amyloid-beta (Ab). It plays a role in Alzheimer s disease. Researchers want to study the effect of sleep on Ab in the brain.

Objective:

To see if sleep affects the amount of waste product removed from the brain.

Eligibility:

Healthy people at least 18 years of age.

Design:

Participants will be screened with a medical history, physical exam, and blood and urine tests. They will answer questions about drug use, psychiatric history, and family history of alcoholism or drug use. Participants will complete an MRI screening questionnaire.

Participants will stay in the clinic overnight two times. On one night they will sleep through the night. On the other night they will be kept awake all night. These overnight visits can happen in any order.

Participants will wear 2 activity monitors, on the wrist and the ankle.

Participants will have positron emission tomography (PET) scans. A small amount of a radioactive chemical will be injected through an intravenous (IV) catheter. Participants will lie on a bed that slides into the scanner. A cap or a special mask may be placed on the participant s head.

Participants will have magnetic resonance imaging (MRI) scans. The MRI scanner is a metal cylinder in a strong magnetic field. Participants will lie on a table that slides into the cylinder. A device called a coil will be placed over the head. Participants will do a task on a computer screen in the scanner.

Participants will have tests of thinking, memory, and attention. They may be interviewed, complete questionnaires, take pen-and-paper or computer tests, and perform simple actions.

DETAILED DESCRIPTION:
Objective:

To assess if there are differences in [18F]florbetaben uptake following the first 120 minutes of its injection (reflecting amyloid-beta or Ab load and/or docked Ab) in subjects during rested wakefulness (RW) after normal sleep compared to wakefulness after 24 hrs of sleep deprivation (SD). Specifically, we hypothesize that during RW after a normal night s sleep there will be less [18F]florbetaben binding measured as distribution volume ratios (DVR) in precuneus relative to cerebellum (reflecting normal brain clearing of Ab overnight) when compared to wakefulness after SD, which would interfere with Ab removal from the brain s interstitial space. Though we will be measuring Ab in whole brain our analysis will focus in precuneus since this is the brain region that shows the higher levels of Ab accumulation in contrast to cerebellum where there is no accumulation of Ab. Therefore, overall Ab load in precuneus (as reflected by [18F]florbetaben DVR) will be lower during RW compared to SD. MRI and 1H-MRS will be used secondarily to assess if there are differences in connectivity, function and neurochemistry in precuneus between RW and SD. Because the rate of CSF production as well as Ab clearance from CSF differs as a function of age the current study will also allow us to assess if the higher Ab brain levels reported in older than in younger individuals reflect greater Ab clearance in younger than older individuals.

Study population:

Two groups consisting of healthy young adults (18 - 40 years of age) and healthy older adults (>40 years of age). Males and females will be included.

Design:

Observational study. We will complete testing in 15 healthy controls in each group for a total of thirty subjects (n=30) to assess the brain uptake of [18F]florbetaben (scan done for 120 minutes following tracer injection). The order of the scans (RW vs SD will be randomized). MRI scans will be obtained either before or after the PET scanning session done following [18F]florbetaben injection.

Outcome measures:

Uptake of [18F]florbetaben in the brain will be measured after RW and after SD. Primary outcomes will be differences in uptake and clearance of [18F]florbetaben in precuneus (reflecting A beta load and/or docked A beta) in subjects after SD compared to after RW as measured with distribution volume ratios using cerebellum as reference region and that clearance of Ab brain (difference between RW and SD) will be greater in younger than in older participants . We hypothesize that Ab load in precuneus [18F]florbetaben DVR) will be higher after SD than RW and that this difference will be larger for younger than older participants. We also predict that older individuals will have higher brain accumulation of Ab than younger ones. In addition we will assess differences in mean water diffusivity in brain, lactate concentration, functional connectivity at rest and functional activation during an attention task between RW and SD conditions. We predict lower fMRI signals in dorsal attention network (DAN) during attention task, lower functional connectivity in the default mode network (DMN), and lower functional connectivity and mean diffusivity for SD than for RW. We further predict higher concentration of lactate, a marker of anaerobic metabolism for SD than for RW. As exploratory analysis we will also assess based on the scans obtained after RW if individuals with higher brain Ab accumulation will have worse cognitive performance on neuropsychological tests than those with low brain Ab.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Male or females.
  2. Young group (18-40 years of age)
  3. Older group (>40 years of age)
  4. Ability to provide written informed consent

EXCLUSION CRITERIA:

1. Pregnant and/or breast feeding. Females of childbearing potential must have negative urine pregnancy test and not be currently breastfeeding. Post-menopausal or surgically sterile (tubal ligation or hysterectomy) females satisfy these criteria.
2. Positive urine drug test for controlled substances (cocaine, methamphetamine, amphetamines, opioids, cannabinoids, benzodiazepines and barbiturates) on each visit involving imaging studies and/or neuropsychological assessment.
3. Head trauma with loss of consciousness for more than 30 minutes as determined by self-report and/or medical history.
4. Subjects with problematic insomnia as determined by self-report (reports having trouble sleeping on most days).
5. Subjects with any of the following: narcolepsy, obstructive sleep apnea (OSA) and/or abnormal sleeping patterns (including but not limited to those who use a CPAP machine, sleeping during the day, using medication to fall asleep, sleeps less than 5 hours per night, night shift workers) as determined by self-report and/or medical history.
6. Use, in the past two weeks, of psychoactive medications (four weeks for fluoxetine) or medications that may affect brain function (including but not limited to opioid analgesics, antidepressants, antipsychotics, benzodiazepines and barbiturates, stimulants) as determined by self-report and/or medical history.
7. Current DSM 5 diagnosis of affective disorder, addiction (other than nicotine of caffeine), PTSD, or schizophrenia.
8. Individuals with cognitive impairment as identified with a score of lower than 24 in the MMSE will be excluded. Further, individuals with impairment sufficient to affect consent capacity even if MMSE is less than 24 will be excluded. We will consult the Ability to Consent Assessment Team (ACAT) in those whose capacity to consent may be questionable.
9. Severe medical problems that can permanently impact brain function (e.g., problems of the CNS; cardiovascular; metabolic, autoimmune, endocrine) as determined by history and clinical exam.
10. Individuals with a medical history of a neurodegenerative disease.
11. Heavy alcohol users. Heavy alcohol users are those individuals who consume more than 5 drinks in one seating (if males) or more than 4 drinks in one seating (if females) more than twice a week will be excluded.
12. Uncontrolled hypertension.
13. Presence of ferromagnetic objects in the body that are contraindicated for MRI of the head (including but not limited to pacemakers or other implanted electrical devices, brain stimulators, some types of dental implants, aneurysm clips, metallic prostheses, permanent eyeliner, implanted delivery pump, or shrapnel fragments) or fear of enclosed spaces as determined by the self-report checklist.
14. Fear of enclosed spaces (claustrophobia) as determined by self-report and medical history.
15. Cannot lie comfortably flat on the back for up to 2 hours in the MRI scanner as determined by self-report.
16. Body weight > 250 kg. This is the upper limit that the bed of the MR scanner can accommodate (clinical exam).
17. Have had previous radiation exposure (from X-rays, PET scans, or other exposure) that, with the exposure from this study, would exceed NIH annual research limits as determined by medical history and physical exam.
18. Study investigators and staff, as well as their superiors, subordinates and immediate family members (adult children, spouses, parents, siblings).

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2016-05-02 (Actual); Primary Completion 2017-01-24 (Actual); Study Completion 2018-07-11 (Actual)

PRIMARY OUTCOMES:
(1) To assess if there are differences in [18F] florbetaben binding(reflecting A load) in subjects after SD compared to RW when measured in the morning. | end of study
  We hypothesize that after SD there will be less clearance of A compared to RW. Therefore, overall brain A load (as reflected by [18F] florbetaben DVRs) will be higher after SD compared to RW.
(2) To assess if there are differences in brain A accumulation during RW and SD and to assess if there are differences in brain Aclearance (comparisons of RW versus SD) between young and older participants. | end of study
  We hypothesize that A brain accumulation will be higher in older than younger participants both during RW and SD and that the differences in brain A (Cross)between RW and SD would be greater in younger than older participants due to greater clearance during SD.

SECONDARY OUTCOMES:
This is an exploratory aim to assess if there are differences in brain function and neurochemistry between RW and SD using MRI and 1H-MRS and determine if the variability on the effects of SD is related to differences in brain glymphatic functio... | end of study
  We hypothesize lower fMRI signals in DAN during a visual attention task, lower functional connectivity in DMN, and lower mean diffusivity in ventral precuneus for SD than for RW. We further hypothesize that higher concentration of lactate, a marker of anaerobic metabolism, on 1H-MRS for SD than for RW. We also hypothesize that brain accumulation (particularly during RW) will be associated with worse cognitive performance on neuropsychological tests.

CONTACTS AND LOCATIONS:
Overall Officials: Dardo G Tomasi, Ph.D., Principal Investigator — National Institute on Alcohol Abuse and Alcoholism (NIAAA)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2016-AA-0059.html